CLINICAL TRIAL: NCT02255006
Title: Effect of Acupuncture to Endothelial Dysfunction Induced by Ischemia-reperfusion Injury Via Adenosine Triphosphate-sensitive Potassium Channels or Prostaglandin Pathway
Brief Title: Effect of Acupuncture to Endothelial Dysfunction Induced by Ischemia-reperfusion Injury
Acronym: AURORAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Weon Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HI13C0580-2
Record Dates: First submitted 2014-09-05; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: volunteer; BMI(25 kg/m2)
MeSH Terms: interventions — Glyburide; Celecoxib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- active acupuncture (Experimental): The participants in this group receive real acupuncture treatment at first. Afterwards crossover study is scheduled to be performed.
  Interventions: Device: Active acupuncture; Drug: Euglucon 5mg; Drug: Celebrex 200mg
- Sham acupuncture (Sham Comparator): The participants in this group receive sham acupuncture treatment at first. afterwards crossover study is scheduled to be performed
  Interventions: Device: Sham acupuncture
- Euglycon (Experimental): Glibenclamide (Euglucon, Roche Pharma) is administered 3 hours before FMD measurement.
  Interventions: Device: Active acupuncture; Drug: Euglucon 5mg
- Celebrex (Experimental): Celebrex(celecoxib, pfizer) 200mg twice daily is administered for 5 days before FMD measurement.
  Interventions: Device: Active acupuncture; Drug: Celebrex 200mg

INTERVENTIONS:
Device: Active acupuncture — Active acupuncture treatment group receive electroacupuncture (EA). For EA treatment, unilateral acupuncture meridian point Pericardium5 (PC5), Pericardium6 (PC6), Stomach36 (ST36), and Stomach37 (ST37) are chosen. Disposable, sterile needles and low frequency electrical stimulator (ES-160, ITO, Japan) are used. Each needle is inserted to the depth of 2cm with a 90 degree angle. Thereafter, needles are connected with the pole and electrical stimulation is applied with 2 Hertz continuous wave current. After FMD measurement, a pneumatic cuff placed above the upper arms is inflated to 200 mmHg for 15 minutes. The cuff is then deflated, and 15 minutes of reperfusion is allowed before FMD measurement again. Acupuncture is performed from after ten minutes of ischemia till end time of reperfusion
  Arms: Celebrex; Euglycon; active acupuncture
Device: Sham acupuncture — For sham intervention, nonacupuncture points are used. Electrical acupuncture is connected but electrical stimulation is not given to sham acupuncture group.
  Volunteers undergo FMD measurement and acupuncture like above methods.
  Arms: Sham acupuncture
Drug: Euglucon 5mg — 8 healthy volunteers are administered 5 mg of glibenclamide (Euglucon, Roche Pharma) 3 hour before FMD measurement. This dosage has previously been shown to be able to completely inhibit forearm KATP channels. With the glibenclamide administration, a 10% dextrose infusion is started and titrated to maintain blood sugar levels between 80 and 120 mg/dL throughout the study period. 3 hours after glibenclamide administration, the subjects undergo FMD measurement before and after ischemia reperfusion injury. During ischemia reperfusion period, active acupuncture treatment is performed for 20 minutes like above method.
  Other Names: Glibenclamide
  Arms: Euglycon; active acupuncture
Drug: Celebrex 200mg — 8 healthy volunteers are administered celecoxib, a selective COX-2 inhibitor, 200 mg twice daily for 5 days. Last dose of celecoxib is administered at morning. Volunteers undergo FMD measurements before and after ischemia reperfusion injury in that morning of last dose of celecoxib. During ischemia reperfusion period, active acupuncture treatment is performed for 20 minutes like above method
  Other Names: Celecoxib
  Arms: Celebrex; active acupuncture

SUMMARY:
Some studies suggest that acupuncture improve flow mediated dilation (FMD) that represents endothelial function, but no study has investigated whether acupuncture protects against ischemia and reperfusion (IR)-induced endothelial dysfunction in humans.

This is a prospective crossover study clinical trial. In the first crossover study, 20 healthy nonsmoking volunteers (25 to 40 years old) will be randomly assigned to acupuncture or control. Endothelium-dependent, FMD of the brachial artery will be measured before and after IR (15 minutes of ischemia at the level of the proximal upper arm followed by 15 minutes of reperfusion). Acupuncture will be performed from 10 minute after ischemia till the end time of reperfusion for 20 minutes. In the second single arm study, 16 volunteers are administered oral 5mg glibenclamide two hours before IR injury (n=8) or selective cox-2 inhibitor celecoxib 200mg twice a day for 5 days to know what mechanism is responsible for acupuncture effect on IR injury. FMD measurements and acupuncture intervention during IR injury are same as above mentioned.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer age 25 to 40 years
* non-smoker

Exclusion Criteria:

* hypertension (>140/90 mmHg), diabetes any cardiovascular disease kidney disease thyroid disease cerebrovascular disease liver disease (bilirubin level >2 mg/dl) pregnancy body mass index >25 kg/m2

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The difference of endothelial function | 4 week
  Endothelial function is measured by brachial flow mediated dilation (FMD). Is there a difference of forearm FMD achieved following ischemia reperfusion injury between acupuncture and control group

SECONDARY OUTCOMES:
The difference of endothelial function | 4 week
  Endothelial function is also measured by brachial flow mediated dilation (FMD). Is the difference of endothelial function mediated by acupuncture hampered by Triphosphate-Sensitive Potassium (KATP) Channels inhibitor glibenclamide or selective cox-2 inhibitor celebrex if acupuncture could improve flow mediated dilation after ischemia reperfusion injury? It is performed for knowing which mechanisms are involved in this improvement if acupuncture could improve flow mediated dilation after ischemia reperfusion injury?

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University Medical Center, Seoul, South Korea